CLINICAL TRIAL: NCT07204080
Title: Phase II Clinical Trial Evaluating the Safety and Efficacy of Fc-Modified Anti-CD154 mAB (TNX-1500) in Kidney Transplant Recipients
Brief Title: (TNX-1500) in Kidney Transplant Recipients
Acronym: TONIX-1500
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ayman Al Jurdi, MD (Other)
Collaborators: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ayman Al Jurdi, MD, Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P-------
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant; Kidney Transplant Failure and Rejection; Immunosuppression; Immunosuppression After Kidney Transplantation
Keywords: Kidney Transplant; New Immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Kidney Transplant Recipient (Experimental)
  Interventions: Drug: TNX-1500; Procedure: Kidney Transplant

INTERVENTIONS:
Drug: TNX-1500 — This is an open-label, single-center, single-arm study to assess the safety and efficacy of TNX-1500, an Fc-modified anti-DF154 mAb in five adult kidney transplant recipients.
Procedure: Kidney Transplant — Kidney Transplant

SUMMARY:
The primary objective is to investigate the safety and efficacy of TNX-1500, an FC-modified anti-CD154 mAb, in five kidney transplant recipients at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 to 75 years of age.
2. Kidney transplant candidates with chronic kidney disease (stage IV or V) or end-stage kidney disease evaluated and listed for transplantation at Massachusetts General Hospital.
3. Recipient of an ABO-compatible, non-human leukocyte antigen (HLA) identical living or deceased donor kidney (de novo or second transplant)
4. Ability to understand the study requirements and provide written informed consent.
5. Epstein-Barr virus (EBV) seropositive

Exclusion Criteria:

1. Recipient seropositive for human immunodeficiency virus (HIV-1), or hepatitis B surface antigen (HBsAg) or core antibody (Anti-HBc); subjects who are seropositive for hepatitis C virus (HCV) are excluded without proof of sustained viral response (SVR) after anti-HCV treatment or spontaneous clearance.
2. Recipient of a kidney from a donor who tests positive for HIV, HBsAg, Anti-HBc, or HCV NAT.
3. Subjects with a severe systemic infection, current or within the 2 weeks prior to screening.
4. Left ventricular ejection fraction < 40% as determined by TTE or clinical evidence of heart failure.
5. Pregnant or nursing (lactating) women confirmed by human chorionic gonadotropin (hCG) laboratory test.
6. Women of childbearing potential (women capable of becoming pregnant) unless using a highly effective method of contraception during dosing and for 24 weeks after study treatment. Highly effective contraception methods include:

   1. Female sterilization (surgical, bilateral oophorectomy with or without hysterectomy), or tubal ligation at least 6 weeks before taking study treatment.
   2. Male sterilization (at least 6 months prior to screening); for female subjects on the study, the vasectomized male partners should be the sole partners for that subject.
   3. Use of injected or implanted hormonal methods of contraception or other hormonal contraception that have comparable efficacy (<1% for example, hormone vaginal ring or placement of a long-acting reversible contraceptives, an intrauterine device, or intrauterine system.
   4. Total abstinence
7. Use of other investigational products or enrollment in another investigational drug study within 30 days prior to screening or 5 half-lives, whichever is longer.
8. Subjects with clinically significant lab abnormalities (>2.5 x the upper limit of normal (ULN) of the following liver function chemistries unless due to, as judged by the investigator, a benign underlying condition:

   1. Alanine aminotransferase (ALT)
   2. Aspartate aminotransferase (AST)
   3. Alkaline phosphatase (ALP)
   4. Bilirubin
   5. Coagulation studies (international normalization ratio (INR), prothrombin time (PT), and partial thromboplastin time (PTT))
9. Any other clinically significant medical condition, active infection, laboratory abnormality, or psychosocial condition (e.g. history of substance use disorder) that would, in the judgement of the investigator, impact the subject's ability to participate in the trial.
10. Subject receives an organ at high risk for delayed graft function, including from a deceased donor after cardiac death (DCD) or a high Kidney Donor Profile Index ≥85%.
11. Presence of pre-existing donor-specific antibodies (DSA) or calculated panel reactive antibodies (cPRA) >20% based upon results within 6 months prior to transplant.
12. Virtual crossmatch (VXM) positive transplant with an MFI >1000 as assessed by routine methodology (Luminex)
13. Cytomegalovirus (CMV) high risk combination: donor positive to recipient negative
14. Multi-organ transplant or tissue recipient.
15. History of malignancy of any organ system, except for localized excised non-melanomatous skin or carcinoma in situ of the cervix
16. Subjects with any of the following: hemoglobin <8 mg/dL, white blood cell ≤2,000/mm3, or platelet count ≤75,000/mm3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events in each subject | 12 Months
  The primary endpoint is the cumulative incidence of all AEs and SAEs in subjects treated with TNX-1500 at 12-months (Day 364, Week 52).
Number of Serious Adverse Events in each subject | 12 Months
  The primary endpoint is the cumulative incidence of all AEs and SAEs in subjects treated with TNX-1500 at 12-months (Day 364, Week 52).

SECONDARY OUTCOMES:
Incidence of Biopsy Proven Acute Rejection | 12 months
  Acute rejection, treatment and outcome biopsy pathology grading (Banff Criteria)
Incidence of treatment for acute rejection | 12 Months
  Acute rejection, treatment and outcome biopsy pathology grading (Banff Criteria)
Incidence of de novo DSA development | Months 1, 3, 6, 9, 12
Incidence of serious opportunistic infections and malignancies | 12 months
  based upon AE/SAE data and available quantitative and qualitative EBV and CMV surveillance data
GFR measurement | 12 months
  Assessment of renal function through the estimated glomerular filtration rate at 12 months post-transplant
Incidence of death | 12 months
Incidence of graft loss | 12 months
Degree of Proteinuria | 12 Months
  Proteinuria by urine protein-to-creatinine ratio
Degree of albuminuria | 12 Months
  Albuminuria by urine microalbumin-to-creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Al Jurdi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No